CLINICAL TRIAL: NCT05532072
Title: Efficacy and Safety Evaluation of Rapamycin Combined With Methylprednisolone in the Treatment of Hyperthyroidism Exophthalmos: A Randomized, Controlled, Multicenter Clinical Trial.
Brief Title: Rapamycin Plus Methylprednisolone Versus Methylprednisolone Alone in Active, Moderate-to-severe Graves' Orbitopathy.
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Collaborators: Beijing Tongren Hospital (Other); Cheloo Hospital (Qingdao), Shandong University (Unknown); Jiangsu Province Hospital with Integration of Chinese and Western Medicine (Unknown); Nanjing First Hospital, Nanjing Medical University (Other); Zhejiang Provincial People's Hospital (Other); Southern Medical University, China (Other); People's Hospital of Xinjiang Uygur Autonomous Region (Other); The Second Affiliated Hospital of Air Force Military Medical University (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: XJTU1AF2021CRF-004
Record Dates: First submitted 2022-04-19; First posted 2022-09-08 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-06

CONDITIONS: Graves Ophthalmopathy
MeSH Terms: conditions — Graves Ophthalmopathy | interventions — Sirolimus; Methylprednisolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- The group of Meprednone combined with Rapamycin (Experimental): The specific dose of methylprednisolone pulse therapy is 500mg / week * 6 + 250mg / week * 6. RAPA has rich experience in the application of renal transplantation, and the recommended maintenance amount for renal transplant patients is 2 mg / day. The efficacy benefits of doses above 2 mg are unclear, and the overall safety of Rapa 2 mg is better than that of patients taking Rapa 5 mg daily. Therefore, based on the clinical experience and clinical research data of RAPA, we would select the dose of Rapamycin as 2mg / day. The experimental group received rapamycin 2 mg/day orally for 24 weeks on the basis of methylprednisolone pulse therapy, and monitor the blood concentration of Rapa at the end of the first week and the end of the 12th week.
  Interventions: Drug: Rapamycin; Drug: Methylprednisolone
- The group of Meprednone alone (Other): The specific dose of methylprednisolone pulse therapy is 500mg / week * 6 + 250mg / week * 6. The effect of methylprednisolone pulse therapy on moderate and severe active Tao has been widely verified in clinical work. EUGOGO will take methylprednisolone pulse therapy as the first-line treatment of moderate and severe active Tao in 2020.
  Interventions: Drug: Methylprednisolone

INTERVENTIONS:
Drug: Rapamycin — Rapamycin plus Methylprednisolone
  Other Names: Sirolimus
  Arms: The group of Meprednone combined with Rapamycin
Drug: Methylprednisolone — Methylprednisolone Alone

SUMMARY:
This study is a randomized, controlled, multi-center clinical study, the purpose is to evaluate the efficacy and safety of rapamycin combined with methylprednisolone in the treatment of moderate to severe active GO.

GO patients with moderate to severe activity were selected as the research objects, and the screening period was 1 week. Eligible and well-informed subjects were randomly assigned 1:1 to the experimental group (rapamycin + methylprednisolone) or the control group (methylprednisolone group). The control group was given methylprednisolone pulse 500 mg/time once a week for 6 weeks + 250 mg/time once a week for 6 weeks, and the experimental group was given rapamycin 2 mg/day orally for 24 weeks on the basis of methylprednisolone pulse therapy. The follow-up period was from 25th to 36th week.

Before treatment, 1 week after treatment, 6 weeks, 12 weeks, 24 weeks, and 36 weeks, visits were conducted to evaluate the improvement and safety evaluation of patients' GO eye activity, severity, and quality of life. At the end of the 1st week and the 12th week, the blood concentration of rapamycin was measured.

DETAILED DESCRIPTION:
Project basis:

Thyroid-associated ophthalmopathy (GO), a vision-threatening autoimmune disease, is the most common extrathyroidal manifestation of Graves disease. At present, GO treatment is still dominated by hormone therapy. From 2010 to 2018, the effective rate of GO hormone shock during moderate to severe activity in our hospital was about 52%. The long-term massive use of hormones can lead to iatrogenic Cushing's syndrome, peptic ulcer, insomnia, delusions, abnormal behavior, pathological fractures, and secondary infections. Therefore, regardless of the disease itself or the treatment method, GO seriously affects the physical and mental health of patients, and optimizing the existing diagnosis and treatment plan has always been a research hotspot in the field. Autoimmunity-induced inflammatory response increased orbital extracellular matrix secretion, and increased fat volume is the cornerstones of the pathogenesis of GO. Previous studies have shown that the PI3K-AKT-mTOR pathway is involved in the synthesis and secretion of extracellular matrix and adipogenesis in orbital fibroblasts. We have demonstrated that RAPA can inhibit orbital collagen and fat deposition in a previous hyperthyroid exophthalmos mouse model. In another small sample (20 patients) study of refractory GD patients, it was also confirmed that methimazole combined with RAPA can effectively reduce thyroid hormone levels, shorten drug withdrawal time, and restore Th17 compared with methimazole alone. /Treg balance. At the same time, there were no adverse reactions in the patients during up to 1 year of follow-up. Therefore, this study intends to carry out large-scale clinical research based on the previous small sample research. A total of 140 patients with GO were enrolled from the endocrinology clinic of our hospital and other hospitals and were randomly divided into two groups. They were treated with methylprednisolone pulse alone and methylprednisolone pulse combined with rapamycin respectively. The clinical and immunological indicators were used to evaluate the effect of RAPA on GO patients. Efficacy and safety, bringing new hope to GO patients.

Research purposes:

To compare the efficacy and safety of rapamycin 2mg/day orally for 24 weeks combined with methylprednisolone pulse therapy and methylprednisolone pulse therapy alone in the treatment of moderate to severe active eye disease.

main target: Rapamycin 2mg/day orally*24 weeks combined with methylprednisolone pulse therapy and methylprednisolone pulse therapy alone in moderate to severe active GO was effective and safe at 24 weeks.

Secondary goals:

1. The effective rate of rapamycin combined with methylprednisolone pulse and methylprednisolone pulse in the treatment of moderate to severe active GO at 36 weeks;
2. At 36 weeks, the recurrence rate of GO in moderate to severe active stage in the treatment of rapamycin combined with methylprednisolone pulse and methylprednisolone pulse therapy;
3. At 24 weeks, the effects of rapamycin and methylprednisolone on GO exophthalmos, CAS, GO-QoL, intraocular pressure, orbital content volume (estimated by MRI), eye cleft width, eye movement, visual acuity, the impact of TRAb.
4. 36 weeks of rapamycin and methylprednisolone shock on GO exophthalmos, CAS, GO-QoL, intraocular pressure, orbital content volume (estimated by MRI), eye cleft width, eye movement, Visual acuity, the effect of TRAb.

Explore goals:

1. To explore the effect of rapamycin combined with methylprednisolone pulse therapy on Th1, Th2, Th17, and other effector T cells and immune regulatory Treg cells in GO patients;
2. To explore the effect of rapamycin combined with methylprednisolone pulse on OF adipogenesis and extracellular matrix secretion.

This study was a multicenter, randomized, controlled study. Study Design: The study was divided into four phases: screening period, dual-drug combination period, monotherapy period, and follow-up period.

Screening period: Experiment-1-0 weeks. According to the inclusion criteria and exclusion criteria, patients with moderate to severe active GO who met the research requirements were selected as the research objects. After obtaining the informed consent of the patients, the research objects were randomly assigned to the control group and the experimental group in a ratio of 1:1. Before formal treatment, peripheral blood was collected for the determination of immune cells and adipogenesis markers.

Dual-drug treatment period: Week 1 to Week 12 of the study. The control group was given methylprednisolone shock control. Experimental group: Based on methylprednisolone pulse therapy, oral administration of rapamycin 2 mg/day was given.

Monotherapy period: From the 13th week to the 24th week of the study, all subjects discontinued methylprednisolone pulse therapy. The experimental group continued to take rapamycin 2 mg orally.

Follow-up period: Week 25 to Week 36. Follow-up observed the improvement of GO eye activity, severity, and quality of life in patients.

Methylprednisolone pulse therapy regimen: Methylprednisolone 500 mg/week*6 weeks + 250 mg/week*6 weeks, the cumulative dose of methylprednisolone is 4.5 g. Proton pump inhibitors and vitamin D and calcium were given as needed during the dual-drug therapy period. Follow-up at Week 0, Week 6, Week 12, Week 24, and Week 36 to assess GO eye disease activity, severity, and GO-QoL improvement. Before the screening, blood was collected at the 2nd visit (1 week + 3 days), the 3rd visit (6 weeks + 3 days), and the 4th visit (12 weeks + 3 days) for safety evaluation. On the 2nd visit (1 weekend + 3 days) and the 4th visit (12 weeks + 3), blood was collected for the determination of rapamycin plasma concentration. After a random assignment at the first visit (0 weeks), the third visit (6 weeks + 3), and the fifth visit (24 weeks + 3 days), samples were collected for mechanism research.

During the study, if the patient developed vision-threatening GO or other conditions, they were required to withdraw from the study.

Research objects:

A total of 140 untreated patients with moderate-to-severe active GO (moderate-severe: 2021 EUGOGO CSS grading criteria; active stage (CAS) ≥ 3), aged 18-70 years.

data analysis: Main objective analysis: Summarize the number and percentage of responding cases at 24 weeks of treatment, using a logistic regression analysis model, with the experimental group as the fixed effect, compare the difference in the compliance rate between groups, and calculate its Odds ratio and 95% confidence interval.

Secondary objective analysis: The logistic regression analysis model was still used for the categorical variables in the secondary objective, and the covariance analysis model was used for continuous variables such as proptosis, GO-QoL, intraocular pressure, and orbital content volume (estimated by MRI). (ANCOVA) analysis.

Safety evaluation: Analysis of safety indicators based on safety analysis set, including adverse events, laboratory tests, physical examination of vital signs (including weight) and electrocardiogram, etc.

Determination of sample size:

The effective rate of MMF combined with methylprednisolone in the treatment of GO was 71%, and we assumed that the effective rate of rapamycin combined with methylprednisolone was 75%. β=0.2, α=0.05, the effective rate of the methylprednisolone treatment group is about 50%, and the effective rate of methylprednisolone combined with the rapamycin treatment group is about 75%. With a preset loss to follow-up rate of 30%, it is planned to enroll 140 patients, 70 in each treatment group.

ELIGIBILITY:
Inclusion Criteria:

1)18-70 years old 2)Clinically diagnosed GO (a. Moderate-severe, b. Active stage)

1. Moderate-severe( CSS Grading Standards for EUGOGO 2021)
2. Active stage (CAS) ≥ 3

Exclusion Criteria:

1. Sight-threatening GO
2. There are obvious abnormalities in laboratory tests: liver damage: ALT and AST ≥ 3 times the upper limit of normal values; kidney damage: serum creatinine ≥ 1.5*ULN; blood routine: hemoglobin < 9g/dl, white blood cell count < 3000/µl or Platelets < 100,000/µl; blood lipids: total cholesterol > 300 mg/dl or triglycerides > 400 mg/dl after lipid-lowering therapy;
3. The patient developed an infection during treatment, requiring intravenous antibiotics, and did not show clinical improvement within 5 days;
4. The subject has a systemic allergic reaction to rapamycin or methylprednisolone;
5. The subject is pregnant during the test;
6. The patient requests to withdraw from the researcher;
7. Investigators believe that they cannot continue to participate in the experiment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Number of participants who responded to treatment as assessed by CAS score, eye cleft width, eye movement, etc. | 24 weeks
  To assess the number of treatment-responsive participants with rapamycin 2 mg/day orally for 24 weeks in combination with pulsed methylprednisolone and pulsed methylprednisolone alone for moderately to severely active GO.
Number of participants with treatment-related adverse events assessed by physical examination, electrocardiogram, and serum biochemical markers. | 24 weeks
  To evaluate the number of participants for treatment-related adverse effects of rapamycin 2 mg/day orally for 24 weeks in combination with pulsed methylprednisolone and pulsed methylprednisolone alone in the treatment of moderately to severely active GO.

SECONDARY OUTCOMES:
Number of participants who responded to treatment as assessed by CAS score, eye cleft width, eye movement, etc. | 36 weeks
  To assess the number of treatment-responsive participants with rapamycin 2 mg/day orally for 24 weeks in combination with pulsed methylprednisolone and pulsed methylprednisolone alone for moderately to severely active GO.
Number of participants with disease recurrence as assessed by CAS score, eye movement, visual acuity, diplopia, etc. | 36 weeks
  The number of participants with disease recurrence in moderately to severely active GO with rapamycin 2 mg/day orally for 24 weeks in combination with pulsed methylprednisolone and pulsed methylprednisolone alone was assessed at 36 weeks.
Antibody titers | 24 weeks
  Effects of rapamycin combined with methylprednisolone pulse therapy and methylprednisolone pulse therapy on TRAb at 24 weeks.
Antibody titers | 36 weeks
  Effects of rapamycin combined with methylprednisolone pulse therapy and methylprednisolone pulse therapy on TRAb at 36 weeks.
GO-QoL Score | 24 weeks
  Effects of rapamycin combined with methylprednisolone pulse therapy and methylprednisolone pulse therapy on GO-QoL Score at 24 weeks.
GO-QoL Score | 36 weeks
  Effects of rapamycin combined with methylprednisolone pulse therapy and methylprednisolone pulse therapy on GO-QoL Score at 36 weeks.
Orbital content volume | 24 weeks
  Effects of rapamycin combined with methylprednisolone pulse therapy and methylprednisolone pulse therapy on orbital content volume at 24 weeks.
Orbital content volume | 36 weeks
  Effects of rapamycin combined with methylprednisolone pulse therapy and methylprednisolone pulse therapy on orbital content volume at 36 weeks.
Intraocular pressure | 24 weeks
  Effects of rapamycin combined with methylprednisolone pulse therapy and methylprednisolone pulse therapy on intraocular pressure at 24 weeks.
Intraocular pressure | 36 weeks
  Effects of rapamycin combined with methylprednisolone pulse therapy and methylprednisolone pulse therapy on intraocular pressure at 36 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Bingyin Shi, Study Chair — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- First Affiliated Hospital of Xian Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol and Clinical Study Report
Supporting Information: Study Protocol, CSR
Time Frame: 2023
Access Criteria: Accepted by author